CLINICAL TRIAL: NCT05078593
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of HLX26 Monoclonal Antibody Injection (Anti LAG-3 Monoclonal Antibody) in Patients With Advanced/Metastatic Solid Tumor or Lymphoma
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of HLX26 Monoclonal Antibody Injection in Patients With Solid Tumor or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX26-001
Record Dates: First submitted 2021-10-13; First posted 2021-10-14 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor, Adult; Lymphoma
Keywords: LAG-3
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX26 (Experimental): The initial dose of HLX26 is 60 mg, and 7 dose levels are designed: 60 mg, 150 mg, 300 mg, 500 mg, 800 mg , 1200mg, and 1600mg(Q3W).
  Interventions: Drug: HLX26

INTERVENTIONS:
Drug: HLX26 — Humanized Anti-Lymphocyte Activation Gene-3 Monoclonal Antibody
  Other Names: Anti-LAG-3 Monoclonal Antibody

SUMMARY:
This study is a first-in-class open-label phase I human clinical study to evaluate the safety and tolerability of HLX26 with escalated doses in the treatment of patients with advanced/metastatic solid tumors or lymphomas.

DETAILED DESCRIPTION:
This study is a first-in-class open-label phase I human clinical study to evaluate the safety and tolerability of HLX26 with escalated doses in the treatment of patients with advanced/metastatic solid tumors or lymphomas. In this study, accelerated titration is combined with a 3 + 3 dose escalation method, and the patients will be given different doses(60mg, 150mg, 300mg, 500mg, 800mg Q3W) of HLX26 intravenously. Observation period of DLT lasts for 3 weeks after the first administration of HLX26.

ELIGIBILITY:
Inclusion Criteria:

1. Have a full understanding of the study content, process, and possible adverse reactions before the study, and sign the informed consent form (ICF); voluntarily participate in the study; be able to complete the study as per protocol requirements;
2. Aged ≥ 18 years at the time of signing the ICF;
3. Patients with histologically or cytologically confirmed advanced malignant solid tumor or lymphoma, who have failed or cannot receive the standard treatment;
4. With at least one measurable lesion according to RECIST V1.1 (for solid tumors) or the Lugano criteria (for lymphomas);
5. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1 at enrollment;
6. Expected survival > 3 months;
7. Have appropriate hematological functions: no blood transfusion or colony stimulating factor therapy (G-CSF) within 14 days before the first administration; absolute neutrophil count ≥ 1500/μL; haemoglobin ≥ 9 g/dL; platelet count ≥ 90,000/μL;
8. Have appropriate coagulation functions: activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; prothrombin time (PT) ≤ 1.5 × ULN; international normalized ratio (INR) ≤ 1.5 × ULN;
9. Have appropriate liver functions: total bilirubin level ≤ 1.5 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 × ULN (AST and ALT ≤ 5 × ULN for patients with known liver metastasis or primary hepatocellular carcinoma);
10. Have appropriate renal functions: blood creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (calculated by Cockcroft-Gault formula);
11. The first administration of the investigational product must be: at least 28 days apart from the previous major surgery, medical device treatment, or local radiotherapy; at least 28 days apart from the previous cytotoxic chemotherapy, immunotherapy, and biological agent therapy; at least 14 days apart from the previous hormone therapy and surgical operation; at least 21 days or 5 half-lives apart from the administration of small molecule targeted drugs, whichever is longer; at least 14 days apart from the traditional Chinese medicine for tumor indications;
12. For patients with hepatocellular carcinoma, Child-Pugh score has to be A;
13. Male and female subjects with child-bearing potential must agree to use at least one highly effective contraception method during the study and within at least 6 months after the last administration of the investigational product.

Exclusion Criteria:

1. The adverse reactions (except alopecia and other adverse reactions determined by the investigator to have no safety risk) of previous anti-tumor therapy have not yet recovered to ≤ grade 1 (CTCAE V5.0);
2. Those who are known to have severe anaphylaxis (grade 4 or greater in CTCAE V5.0) to macromolecular protein preparations/monoclonal antibodies or to any component of the investigational product;
3. Patients with any of the following unstable or poorly controlled diseases:1)Active systemic infectious diseases requiring intravenous antibiotics within 2 weeks before the first administration of the investigational product;2)Any poorly-controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited to: (1) NYHA Class II or greater cardiac failure or left ventricular ejection fraction (LVEF) < 50%; (2) unstable angina pectoris; (3) myocardial infarction and cerebral infarction within 6 months, (4) clinically significant supraventricular or ventricular arrhythmia without clinical intervention or poorly controlled after clinical intervention;3)Other chronic diseases which, in the opinion of the investigator, may compromise the safety of the patient or the integrity of the study;
4. Assessed as unsuitable for inclusion by the investigator, due to brain metastases, spinal cord compression, or cancerous meningitis with clinical symptoms, or uncontrolled brain or spinal cord metastases that have been evidenced;
5. Previous grade 3 or greater irAEs in immunotherapy;
6. Have had other malignant tumors within 5 years before enrollment, except: (a) those with cured cervical carcinoma in situ or non-melanoma skin cancer; (b) those with cured second primary cancer without recurrence within 5 years; (c) those with double primary cancers believed to be able to benefit from this study; (d) those whose metastasis has been clearly excluded from a certain primary tumor source; (e) those who have received anti-LAG-3 antibody therapy;
7. Have active autoimmune diseases (including but not limited to the following diseases or syndromes, such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism), except: vitiligo or cured childhood asthma/allergy that does not need any intervention in adulthood, autoimmune mediated hypothyroidism treated with stable dose of thyroid replacement hormone, and type I diabetes treated with stable dose of insulin; those in a stable condition and requiring no systemic immunosuppressant therapy (including corticosteroid hormone) are allowed to be enrolled;
8. Have received systemic corticosteroids (prednisone > 10 mg/d or equivalent dose of similar drug) or other immunosuppressants within 14 days before the first administration; Except: patients treated with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; those with short term use of corticosteroids for prophylaxis, such as contrast agents;
9. Patients in pregnancy [confirmed by serum beta-human chorionic gonadotropin (ß-HCG) test] or breastfeeding;
10. With a history of immunodeficiency, including human immunodeficiency virus (HIV)-positive or other acquired or congenital immunodeficiencies, or a history of organ transplantation;
11. Patients with active HBV or HCV infection (HBV DNA ≥ 104 copies/mL or positive HCV RNA);
12. Have received live vaccines within 30 days prior to the first administration;
13. Patients whose medical history or any other evidence suggests that participation in the study may confuse the results, or subjects for whom the investigator believes the study is not in their best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
The Dose-Limiting Toxicity (DLT) of HLX26 within 3 weeks after the first Administration in patients with Advanced/Metastatic Solid Tumors or Lymphomas | from day1 to day 21
  DLT
The Maximum Tolerated Dose (MTD) of HLX26 within 3 weeks after the first Administration in patients with Advanced/Metastatic Solid | from day1 to day 21
  MTD

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu R, Jing H, Chen Y, Gao S, Zhang J, Cao X, Li K, Liu Y, Meng M, Chen C, Sun C, Yu H, Wang Q, Li J, Wu Y, Zhang J. Phase I Studies of HLX26, A Novel Anti-LAG-3 Antibody, Monotherapy or Combination Therapy in Patients with Advanced Solid Tumors. BioDrugs. 2026 Jan 15. doi: 10.1007/s40259-025-00751-z. Online ahead of print. PMID 41538111